CLINICAL TRIAL: NCT00988000
Title: Telephone Consultations for New Patients Being Referred to a Specialist Respiratory Outpatient Clinic
Brief Title: Initial Specialist Telephone Consultation With New Patients in Secondary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: The Dunhill Medical Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NHLICX07Q060519
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Respiratory Diseases
Keywords: outpatients
MeSH Terms: conditions — Respiratory Tract Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Agree to the alternative study invitation (Other): Agree with alternative of telephone consultation (instead of face to face) offered as an initial consultation to new referrals
  Interventions: Other: telephone consultation
- Decline the alternative study invitation (Other): Decline, no respond to the alternative of telephone consultation
  Interventions: Other: No intervention
- Comparator (Other): Choose and book
  Interventions: Other: No intervention

INTERVENTIONS:
Other: telephone consultation — alternative to face to face consultation for new referrals
  Arms: Agree to the alternative study invitation
Other: No intervention — no alternative to face to face consultation
  Arms: Comparator; Decline the alternative study invitation

SUMMARY:
Consultations with patients by hospital consultants are organised today in a manner which is barely dissimilar from that offered 30 or 40 years ago. Whilst some attempts to improve this process, such as Choose and Book, shorter waiting times and patients' receiving a copy of the correspondence sent to their general practitioner (GP) have improved the situation, there has been little radical change and little thought given to the patient experience.

The investigators wish to investigate whether patients' experience of attending respiratory outpatient clinics can be improved by a pre-clinic telephone call with a specialist thereby reducing the number of attendances at the hospital for appointments and investigations and improving overall patient satisfaction.

DETAILED DESCRIPTION:
This study will investigate whether taking a new patient's history over the telephone permits better selection and arrangement of investigations prior to or synchronous with the first face to face consultation, with the potential to reduce the number of visits the patient has to make to the hospital.

Patients will be offered an initial telephone consultation by post and may opt-in or out of the study. Those having a telephone consultation would have this booked for a specific time and date and the patient would be sent an appropriate information leaflet regarding this. After the telephone consultation patients receive a summary of the consultation and details of any investigations and appointments booked by the research nurse. Patients who did not respond to the initial invitation letter within seven days or who declined to participate would be sent a routine appointment. All patients would asked to complete the MISS-21 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* All new adult general respiratory referrals from primary care

Exclusion Criteria:

* Follow-up patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor MR Partridge, MD FRCP, Principal Investigator — Imperial College London
Locations (1):
- Imperial College at Charing Cross campus, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients' who attending respiratory outpatient clinics
Groups:
- Agree to Alternative Study Invitation: Patients Respond to study invitation - agree to alternative consultation
- Declined the Alternative Study Invitation: Patients respond to study invitation - declined/ non-responders for the invitation
- Comparator: Patients - choose and book
Period: Overall Study
Arm/Group | Agree to Alternative Study Invitation | Declined the Alternative Study Invitation | Comparator
Started | 49 | 51 | 57
Completed | 49 | 51 | 57
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Respond to Study Invitation - Agree to Alternative Consultatio: participants agreed to have an alternative consultation i.e. telephone consultation for their first hospital appointment
- Respond to Study Invitation - Declined/ Non-responders: Participants declined or did not respond to the invitation to participate in the study
- Comparator - Choose and Book: participants in this group booked their appointment through the choose and book system
- Total: Total of all reporting groups
Arm/Group | Respond to Study Invitation - Agree to Alternative Consultatio | Respond to Study Invitation - Declined/ Non-responders | Comparator - Choose and Book | Total
Number analyzed (Participants) | 49 | 51 | 57 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (13.7) | 57.4 (16.7) | 50.9 (17.0) | 56.7 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 28 | 83
  Male | 22 | 23 | 29 | 74
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 49 | 51 | 57 | 157

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction of the Alternative Consultation
Description: Patient Satisfaction assessed by MISS scale, Medical interview satisfaction score. The score 0-7, 0 means dissatisfaction, higher scores indicate higher satisfaction.
Time Frame: First clinic appointment (Month 0) and Follow-up appointment (6 months
Population: Incomplete data and those that had an alternative consultation did not need a follow up appointment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Agree to the Alternative Consultation: Patients respond to study invitation and agree
- Declined the Alternative Study Invitation: Declined/non-responders for the invitation
- Comparator: Patients choose and book
Arm/Group | Agree to the Alternative Consultation | Declined the Alternative Study Invitation | Comparator
Number analyzed (Participants) | 44 | 29 | 41
score on a scale
  first clinic appointment | 5.85 (0.73) | 5.67 (0.68) | 5.26 (0.70)
  follow-up appointment: number analyzed (Participants) | 0 | 17 | 17
  follow-up appointment |  | 5.47 (0.53) | 5.36 (0.98)

2. Secondary Outcome: Number of Required Investigations
Description: reduction in number of required investigations
Time Frame: 0-6 months
Measure: Number; unit: number of investigation
Groups:
- Agree to the Alternative Study Invitation: Patients respond to study invitation and agree
- Declined the Alternative Study Invitation: Declined/ non-responders to the alternative study invitation
Arm/Group | Agree to the Alternative Study Invitation | Declined the Alternative Study Invitation | Comparator
Number analyzed (Participants) | 49 | 51 | 57
number of investigation
  Planned investigations | 147 | 117 | 128
  Completed investigations | 145 | 105 | 116

ADVERSE EVENTS:
Time Frame: 10 month
Groups:
- Agree to Alternative Study Invitation: Patients agree to alternative study invitation
- Declined the Alternative Study Invitation: Patients who declined/ non-responders to alternative study invitation
Arm/Group | Agree to Alternative Study Invitation | Declined the Alternative Study Invitation | Comparator
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51 | 0/57
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes